CLINICAL TRIAL: NCT04404361
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Multicenter Study of Pacritinib Plus Standard of Care Versus Placebo and Standard of Care in Hospitalized Patients With Severe COVID-19 With or Without Cancer
Brief Title: PRE-VENT Study in Hospitalized Patients With Severe COVID-19 With or Without Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: decision to close enrollment early
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAC319
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: COVID19; COVID-19; COVID
Keywords: COVID19; COVID-19; COVID
MeSH Terms: conditions — COVID-19 | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Janus Kinase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pacritinib and SOC (Experimental): Pacritinib 400 mg once daily [QD] on Day 1, then 200 mg twice daily [BID] from Day 2 to Day 14) + SOC
  Interventions: Drug: Pacritinib
- Placebo and SOC (Placebo Comparator): 4 capsules once daily [QD] on Day 1, then 2 capsules twice daily [BID] from Day 2 to Day 14) + SOC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pacritinib — 100 mg capsules
  Other Names: SB1518; Oral Jak Inhibitor; Oral Irak inhibitor; Oral Csf1 inhibitor
  Arms: Pacritinib and SOC
Drug: Placebo — Placebo capsules matching pacritinib 100 mg capsules
  Arms: Placebo and SOC

SUMMARY:
This is a Phase 2 randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of pacritinib in hospitalized patients with severe COVID-19 with or without cancer.

DETAILED DESCRIPTION:
This is a Phase 2 randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of pacritinib in hospitalized patients with severe COVID-19 with or without cancer. Severe COVID-19 is defined as confirmed disease in patients who are hospitalized with hypoxia (blood oxygen saturation [SpO2] ≤93% on room air at sea level), respiratory rate >30, arterial oxygen partial pressure [PaO2]/ fraction of inspired oxygen [FiO2] <300, or lung infiltrates >50% but do not require IMV.

Patients will be randomized 1:1 to receive pacritinib (400 mg once daily [QD] on Day 1, then 200 mg twice daily [BID] from Day 2 to Day 14) + SOC or placebo + SOC.

Assigned treatment will continue for up to Day 14 or until the patient experiences intolerable adverse events (AEs), withdraws consent, or initiates another investigational therapy or until the study is terminated. Assigned therapy may be given for an additional 7 days (for a total of 21 days) with the approval of the Medical Monitor if, in the opinion of the investigator, the patient's clinical signs and symptoms are improving and the potential benefit outweighs the potential risk.In the event of hospital discharge, patients will complete treatment with the assigned therapy as an outpatient.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized or will be hospitalized prior to randomization for the treatment of severe COVID-19 with SARS-CoV-2 infection confirmed by either a) a positive reverse transcriptase polymerase chain reaction (RT PCR) or b) an antigen-based test from any respiratory, nasopharyngeal, saliva, blood, or stool specimen at Screening or documented within 1 week prior to the start of Screening (Severe COVID-19 is defined as confirmed disease in patients who are hospitalized with hypoxia [SpO2 ≤93% on room air], respiratory rate >30, PaO2/FiO2 <300, but do not require IMV).
2. Age ≥ 18 years
3. Platelet count ≥ 50,000/µL
4. If fertile, willing to use effective birth control methods during the study
5. Provision of informed consent within 96 hours after hospitalization

Exclusion Criteria:

1. In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
2. Currently intubated or intubated between screening and randomization
3. Suspected active uncontrolled bacterial, fungal, viral, or other infection (besides COVID 19)
4. Prior allogenic hematopoietic stem cell transplantation
5. Active lung cancer or history of lung cancer within the past 12 months
6. Any active grade 2 or higher hemorrhage
7. Any active gastrointestinal or metabolic condition that could interfere with absorption of oral medication
8. Uncontrolled intercurrent illness that, in the judgment of the treating physician, would limit compliance with study requirements
9. Known seropositivity for human immunodeficiency virus with cluster of differentiation 4 (CD4) count < 200/mm3 within 3 months prior to randomization
10. Pregnant or breastfeeding, or positive pregnancy test in a pre-dose examination
11. Concurrent enrollment in another interventional trial (investigational COVID-19 antiviral studies are permitted)
12. Serum creatinine > 2.5 mg/dL
13. Total bilirubin > 4× the upper limit of normal
14. QT corrected by the Fridericia method (QTcF) prolongation > 480 msec
15. Known history of New York Heart Association Class II, III, or IV congestive heart failure prior to hospital admission
16. Known allergic reaction to any Janus kinase 2 (JAK2) inhibitor
17. Exposure to any JAK2 inhibitor within 28 days
18. Currently receiving a strong CYP3A4 inhibitor or strong P450 inducer (Appendix 1 and Appendix 2, respectively) and unable to stop the medication prior to the first dose of study drug and throughout the duration of study drug administration
19. Treatment with cytoreductive chemotherapy administered within 14 days prior to randomization
20. Administration of an IL 1 or IL 6 blocking immunomodulatory agent (such as tocilizumab, canakinumab, sarilumab, anakinra) within 48 hours prior to randomization
21. Currently receiving therapeutic anticoagulation or anti platelet medication and unable to stop the medication prior to randomization. Prophylactic anticoagulation therapy or aspirin (≤ 100mg) are permitted.
22. Unable to ingest capsules or tablets at randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - St. Jude Hospital Yorba Linda dba St. Joseph Heritage Healthcare, Orange, California
  - Ascension St. Vincent's Riverside Hospital, Jacksonville, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - St. Vincent Medical Group, Inc, Indianapolis, Indiana
  - St. Agnes Healthcare, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Ascension Providence Hospital - Novi Campus, Novi, Michigan
  - Providence Cancer Institute, Southfield, Michigan
  - Atlantic Melanoma Center, Morristown, New Jersey
  - Overlook Medical Center, Morristown, New Jersey
  - Chilton Medical Center, Pompton Plains, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - The Carl and Edyth Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - St. John Medical Center, Tulsa, Oklahoma
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Ascension St. Francis Hospital, Milwaukee, Wisconsin
  - Ascension All Saints, Racine, Wisconsin

REFERENCES:
- [Derived] Cafardi J, Miller C, Terebelo H, Tewell C, Benzaquen S, Park D, Egan P, Lebovic D, Pettit K, Whitman E, Tremblay D, Feld J, Buckley S, Roman-Torres K, Smith J, Craig A, Mascarenhas J. Efficacy and Safety of Pacritinib vs Placebo for Patients With Severe COVID-19: A Phase 2 Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2242918. doi: 10.1001/jamanetworkopen.2022.42918. PMID 36469321

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pacritinib and SOC | Placebo and SOC
Started | 99 | 101
Completed | 68 (Patients who completed the study through 30 days after last dose of study treatment) | 80 (Patients who completed the study through 30 days after last dose of study treatment)
Not Completed | 31 | 21
Not completed — Death | 12 | 12
Not completed — Withdrawal by Subject | 13 | 5
Not completed — Lost to Follow-up | 6 | 3
Not completed — patient hospitalized and was nonverbal at the end of the study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pacritinib and SOC | Placebo and SOC | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Median (Full Range); unit: years] | 60.0 [19 to 87] | 59.0 [28 to 94] | 60.0 [19 to 94]
Age, Customized [Count of Participants; unit: Participants] — Age groups <60 years and ≥60 years
  Participants
    Age group: <60 years | 48 | 51 | 99
    Age group: ≥60 years | 51 | 50 | 101
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 37 | 80
  Male | 56 | 64 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 14 | 27
  Not Hispanic or Latino | 79 | 81 | 160
  Unknown or Not Reported | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 17 | 19 | 36
  White | 74 | 72 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 99 | 101 | 200

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression to IMV and/or ECMO or Death
Description: The percentage is calculated as the number of patients who progress to IMV/ECMO or death divided by the total number of patients in the ITT population (n/N * 100).
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib and SOC | Placebo and SOC
Number analyzed (Participants) | 99 | 101
Participants | 26 | 25
Statistical Analysis 1: Comparison: Pacritinib and SOC vs Placebo and SOC; Test type: Superiority; p = 0.8516, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by age (<60 years versus ≥60 years) and 7-point clinical status scale (baseline 3 or 4 versus 5); Risk Difference (RD) = 1.51, 95% CI 2-sided [-10.55 to 13.53]

2. Secondary Outcome: The Number of Ventilator-Free Days
Description: the number of days that patients are alive and not intubated, from randomization to Day 28
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pacritinib and SOC | Placebo and SOC
Number analyzed (Participants) | 99 | 101
days | 22.1 (10.2) | 22.6 (9.35)
Statistical Analysis 1: Comparison: Pacritinib and SOC vs Placebo and SOC; Test type: Superiority; p = 0.7494, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: The Mortality Rate at Day 28
Description: the number of patients with outcome of death during the 28 days following randomization
Time Frame: Baseline to Day 28
Measure: Number (95% Confidence Interval); unit: % of patients with outcome of death /D28
Arm/Group | Pacritinib and SOC | Placebo and SOC
Number analyzed (Participants) | 99 | 101
% of patients with outcome of death /D28 | 10.1 [5.0 to 17.8] | 7.9 [3.5 to 15.0]
Statistical Analysis 1: Comparison: Pacritinib and SOC vs Placebo and SOC; Test type: Superiority; p = 0.6323, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.46 to 3.58] — OR from a CMH test stratified by randomization stratification factors age (<60 years versus ≥60 years) and 7-point clinical status scale (baseline 3 or 4 versus 5) as entered in the IXRS

4. Secondary Outcome: The Mortality Rate at Day 15
Description: the number of patients with outcome of death in the 15 days following randomization
Time Frame: Baseline to Day 15
Measure: Number (95% Confidence Interval); unit: % of patients with outcome of death /D15
Arm/Group | Pacritinib and SOC | Placebo and SOC
Number analyzed (Participants) | 99 | 101
% of patients with outcome of death /D15 | 5.1 [1.7 to 11.4] | 4.0 [1.1 to 9.8]
Statistical Analysis 1: Comparison: Pacritinib and SOC vs Placebo and SOC; Test type: Superiority; p = 0.7541, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.31 to 4.96] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: The Time to Improvement by at Least 2 Points Relative to Baseline on the 7-point Ordinal Scale of Clinical Status
Description: Time to Improvement (days) = Date of improvement - Date of randomization + 1. Date of Improvement was defined as the time to first ordinal scale assessment 2 points or more lower than the baseline clinical status assessment.
Time Frame: Baseline, Day 8, 15, 22, and 28.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pacritinib and SOC | Placebo and SOC
Number analyzed (Participants) | 99 | 101
days | 9.0 [8.0 to 10.0] | 9.0 [7.0 to 11.0]
Statistical Analysis 1: Comparison: Pacritinib and SOC vs Placebo and SOC; Test type: Superiority; p = 0.5666, Log Rank — log-rank test stratified by randomization stratification factors age (<60 years versus ≥60 years) and 7-point clinical status scale (baseline 3 or 4 versus 5) as entered in the IXRS; stratified by randomization stratification factors age (<60 years versus ≥60 years) and 7-point clinical status scale (baseline 3 or 4 versus 5); Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.79 to 1.53] — estimated using a stratified Cox proportional hazards model stratified by randomization stratification factors age (<60 years versus ≥60 years) and 7-point clinical status scale (baseline 3 or 4 versus 5)

6. Secondary Outcome: The Clinical Status as Assessed by the 7-point Ordinal Scale of Clinical Status at Days 8, 15, 22, and 28
Description: Clinical status assessment based on the adapted scale from Cao et al. The patient CS is summarized by study visit.
  STATUS:
  1. not hospitalized with resumption of normal activities;
  2. not hospitalized but unable to resume normal activities;
  3. hospitalization, not requiring supplemental oxygen;
  4. hospitalization, requiring supplemental oxygen not meeting the criteria for categories 5 or 6;
  5. hospitalization, on non-invasive positive pressure ventilation or high-flow nasal cannula;
  6. hospitalization, requiring IMV and/or ECMO;
  7. death.
Time Frame: Baseline, Day 8, 15, 22, 28
Measure: Number; unit: participants
Arm/Group | Pacritinib and SOC | Placebo and SOC
Number analyzed (Participants) | 99 | 101
participants
  Day 8 : Clinical status 1 | 15 | 11
  Day 8 : Clinical status 2 | 23 | 37
  Day 8 : Clinical status 3 | 5 | 3
  Day 8 : Clinical status 4 | 20 | 11
  Day 8 : Clinical status 5 | 15 | 20
  Day 8 : Clinical status 6 | 9 | 14
  Day 8 : Clinical status 7 | 0 | 1
  Day 8 : Clinical status Missing | 12 | 4
  Day 15: Clinical status 1 | 19 | 17
  Day 15: Clinical status 2 | 43 | 47
  Day 15: Clinical status 3 | 1 | 1
  Day 15: Clinical status 4 | 2 | 8
  Day 15: Clinical status 5 | 5 | 2
  Day 15: Clinical status 6 | 10 | 16
  Day 15: Clinical status 7 | 0 | 2
  Day 15: Clinical status Missing | 19 | 8
  Day 22: Clinical status 1 | 27 | 24
  Day 22: Clinical status 2 | 36 | 48
  Day 22: Clinical status 3 | 1 | 0
  Day 22: Clinical status 4 | 0 | 1
  Day 22: Clinical status 5 | 4 | 1
  Day 22: Clinical status 6 | 7 | 12
  Day 22: Clinical status 7 | 3 | 1
  Day 22: Clinical status Missing | 21 | 14
  Day 28: Clinical status 1 | 31 | 30
  Day 28: Clinical status 2 | 32 | 42
  Day 28: Clinical status 3 | 0 | 0
  Day 28: Clinical status 4 | 3 | 2
  Day 28: Clinical status 5 | 2 | 1
  Day 28: Clinical status 6 | 6 | 10
  Day 28: Clinical status 7 | 0 | 1
  Day 28: Clinical status Missing | 25 | 15

7. Secondary Outcome: The Rate of Use of Immunomodulatory Agents as Treatment for COVID-19
Description: the proportion of patients reporting use of medications such as corticosteroids, tocilizumab, anakinra, or eculizumab as treatment for COVID-19, during 28 days following randomization
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib and SOC | Placebo and SOC
Number analyzed (Participants) | 99 | 101
Participants | 97 | 96
Statistical Analysis 1: Comparison: Pacritinib and SOC vs Placebo and SOC; Test type: Superiority; p = 0.2722, Chi-squared; Odds Ratio (OR) = 2.46, 95% CI 2-sided [0.47 to 12.93]

ADVERSE EVENTS:
Time Frame: Daily (Days 2 through 28), End of Treatment (for inpatients only), Day of hospital discharge, Weekly outpatient assessment (to evaluate daily AEs), 30-day Post End of Treatment. AE data were collected from the time of randomization through 30 days following the last dose of pacritinib/placebo.
Description: regular investigator assessment
  3 patients randomized to PAC but received the Placebo + SOC, the randomized treatment did not match with the actual treatment received. Because this is a safety summary the Safety population summarizes the information according to the actual treatment received and not the treatment that was assigned (randomized).
Arm/Group | Pacritinib and SOC | Placebo and SOC
All-Cause Mortality (participants affected / at risk) | 12/96 | 12/101
Serious Adverse Events (participants affected / at risk) | 20/96 | 33/101
Other Adverse Events (participants affected / at risk) | 74/96 | 79/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacritinib and SOC (N=96) | Placebo and SOC (N=101)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 15 (15)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (8)
septic shock (Infections and infestations) | 2 (2) | 6 (6)
acute kidney injury (Renal and urinary disorders) | 3 (3) | 3 (3)
cardiac arrest (Cardiac disorders) | 1 (1) | 3 (3)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
hypotension (Cardiac disorders) | 2 (2) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacritinib and SOC (N=96) | Placebo and SOC (N=101)
Alanine aminotransferase increased (Hepatobiliary disorders) | 15 (17) | 17 (19)
anaemia (Blood and lymphatic system disorders) | 12 (12) | 18 (18)
bradycardia (Cardiac disorders) | 15 (15) | 11 (11)
constipation (Gastrointestinal disorders) | 12 (12) | 13 (13)
hypokalaemia (Metabolism and nutrition disorders) | 12 (12) | 12 (17)
hyperkalaemia (Metabolism and nutrition disorders) | 9 (9) | 11 (17)
acute kidney injury (Renal and urinary disorders) | 9 (15) | 7 (7)
hypotension (Cardiac disorders) | 8 (9) | 8 (13)
diarrhoea (Gastrointestinal disorders) | 12 (12) | 4 (4)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 9 (9) | 6 (6)
hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 11 (11)
hypertension (Cardiac disorders) | 5 (5) | 8 (8)
hypocalcaemia (Metabolism and nutrition disorders) | 4 (8) | 8 (12)
insomnia (Nervous system disorders) | 6 (6) | 6 (6)
atrial fibrillation (Cardiac disorders) | 5 (5) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 4 (4)
nausea (General disorders) | 4 (4) | 6 (6)
anxiety (Psychiatric disorders) | 6 (7) | 3 (3)
agitation (Psychiatric disorders) | 3 (3) | 5 (5)
thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
encephalopathy (Nervous system disorders) | 1 (1) | 5 (5)
epistaxis (General disorders) | 2 (2) | 5 (5)
headache (Nervous system disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT04404361/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT04404361/SAP_001.pdf